CLINICAL TRIAL: NCT05224882
Title: Oral Manifestations Of Pediatric Cancer Patients Receiving Chemotherapy And Dental Awareness Among Parents
Brief Title: Chemotherapy Oral Manifestations and Dental Awareness Among Parents
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Mohammed Al-Sayed, Principal Investigator, Cairo University
Other Study IDs: Chemotherapy manifestations
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Mucositis Oral; Chemotherapy Effect
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevention of oral illnesses in children and adolescents undergoing oncological treatment is critical, because oral lesions caused by this therapy significantly exacerbate the clinical condition and increase the risk of infection, as well as making it harder to perform required dental procedures when needed .

"The key to success in maintaining a healthy oral cavity during therapy is patient compliance. The child and the parents should be educated regarding the possible acute side effects." Pediatric cancer patients may have a lower quality of life if they have poor dental health. Preventing and treating pre-existing oral illnesses is critical to reduce problems in these people.

It is critical to raise awareness of the benefits of proper oral health so that this understanding becomes a positive attitude, reducing the discomfort of these children.

The American Academy of Pediatric Dentistry (AAPD) recommends pediatric oncology/hematology that Pediatric dentists must be involved in the treatment process from the moment cancer is diagnosed. This should be carried out by having a preventive and dental care plan developed based on the patient's needs before any cancer treatment is initiated.

The aim of the study is primarily to report oral complications and manifestations during chemotherapy treatment in pediatric cancer patients and raise the awareness of their parents on these manifestations thus proper interventions can be carried out to prevent more serious problems.

DETAILED DESCRIPTION:
Childhood cancer is defined here as cancer in children aged 0-14 years and it only accounts for a small portion of the worldwide cancer burden .with an estimated 13.7 million additional cases of cancer in children globally between 2020 and 2050.

Childhood malignancies continue to be a leading source of morbidity and death in children. Cancer is the leading cause of disease-related mortality among children in developed, high-income countries, such as the United States.

With advances in healthcare access and a drop in communicable disease mortality, paediatric cancer is projected to become a significant cause of death even in developing, low- and middle-income nations. Furthermore, because children make up a significant proportion of the population in these countries, the scope of the problem is exacerbated, potentially resulting in a greater burden of childhood malignancy for the healthcare system to address.

Leukaemia accounted for the greatest share of classified childhood cancer burden globally, followed by brain and nervous system cancers.

The Children's Cancer Hospital in Egypt (CCHE) is the country's largest paediatric cancer hospital, enrolling about 3000 children under the age of 18 annually, accounting for an estimated 50% of juvenile cancer cases in a country with a population of around 100,000,000.

The primary mode of treatment for malignancies in children is antineoplastic chemotherapy, either alone or in conjunction with surgery and/or radiation according to the type of neoplasm.

Childhood cancers tend to respond well to chemotherapy as they are fast-growing and thus more susceptible to chemotherapy.This mechanism of treatment usually associated with severe side effects. Moreover, general adverse events that are common among patients treated by chemotherapy include reduced immunity, pancytopenia, muscle atrophy, skin manifestations, hair loss and others.

Chemotherapy includes the administration of injectable pharmaceuticals, which suppresses the immunity .Approximately 15 days after the chemotherapy session, patients usually show immunosuppression. As a result, any change in the integrity of the oral mucosa, carious processes, or outbreaks of odontogenic infection pose a significant risk for the development of additional oral and systemic illnesses.

Complications might be acute (occurring during therapy) or chronic (occurring after therapy) (developing months to years after therapy) Oral problems result from both direct injury to oral tissues as a result of chemotherapy and indirect damage as a result of regional or systemic toxicity.

One of the most common adverse effects of chemotherapy antineoplastic therapy is oral mucositis, which appears as mucosal inflammation followed by tissue degradation caused by chemotherapeutic drug stomatotoxicity. Oral mucositis occurs five to seven days after the start of antineoplastic therapy and lasts for the duration of the treatment.

Also, infections (viral- fungal- bacterial), salivary gland dysfunction, taste impairment, and discomfort are the most frequent oral problems associated with cancer treatments. Secondary problems such as dehydration, dysgeusia, and malnutrition might result from these issues. The mouth cavity can potentially be a source of systemic infection in myelosuppressed cancer patients. Fungal infections and ulceration can be observed with patient on chemotherapy.

Parents of children receiving cancer treatment, particularly chemotherapy, who are in a phase of acute immunosuppression usually neglect dental care. The parents are more concerned about the concurrent disease than the dental care of their kid, as they appeared anxious when presented with a cancer diagnosis, and they inquired about the impact of oral hygiene on cancer therapy and may not see it as a high priority.

ELIGIBILITY:
Inclusion Criteria:

* Children between the age of 1 -14years.
* Children receiving chemotherapy for hematological cancer or solid tumors.
* Parents who are able to understand the aim of the study and willing to participate in the study.

Exclusion Criteria:

* Children previously received radiotherapy on head and neck region.
* Children suffering from oral cancer.
* Children presented with other oral disorders such as leukoplakia.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will be carried out at the pediatric clinic of the National Cancer Institute ,Egypt.
  Pediatric patients and their parents at the pediatric clinic will be screened until the target population is achieved. The pediatric patients will be subjected to thorough examination. Once the patient and the parent are potentially eligible for this study, the principal investigator will explain the study and ascertain the patient's and the parents' interest. The legal guardian provides written informed consent for participation in the study.
Sampling Method: Probability Sample
Enrollment: 441 (Estimated)
Dates: Start 2023-08-12 (Estimated); Primary Completion 2023-11-27 (Estimated); Study Completion 2024-01-25 (Estimated)

PRIMARY OUTCOMES:
The assessment of the prevalence of oral adverse events induced by chemotherapy in pediatric cancer patients . | Baseline
  Patients will be examined for oral manifestations at the first visit together with intra oral photos will be taken for the patients included in the study.
  Voice ,swallow ,tongue, saliva, mucous membrane**, gingiva ,teeth will be measured by Oral Assessment Guide by the principal investigator .
  **If oral mucositis is present it will be staged according to the World Health Organization Scale (WHO Oral Toxicity Scale) by the principal investigator.

SECONDARY OUTCOMES:
Assessment of dental awareness among parents of pediatric cancer patients . | Baseline
  Questionnaire (structured questionnaire that is developed and validated by Gupta et al., 2016) Parents of the pediatric cancer patients participating in the study will complete the "Parental dental Awareness Questionnaire" to assess their awareness.

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Bahgat, Professor, Study Chair — Professor of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Cairo University.

IPD SHARING:
Plan to Share IPD: Undecided